CLINICAL TRIAL: NCT04036162
Title: Spatial and Dynamic Characterization of Brain Activity for Language and Posture (Verticality) During Normal Aging. Magnetoencephalography (MEG) Study (MEG-AGING)
Acronym: MEG-AGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.294; 2019-A01065-52 (Other: ANSM ID RCB)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
Keywords: Aging; Task-Positive Network (TPN); Task-Negative Network (TNN); MagnetoEncephaloGraphy (MEG); Verticality; Language; Hemispheric asymmetry
MeSH Terms: conditions — Language

STUDY DESIGN:
Intervention Model Description: Right-handed healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young group (Experimental): Young Right-handed healthy volunteers
  Interventions: Behavioral: Cognitive tasks
- Aged group (Experimental): Aged Right-handed healthy volunteers
  Interventions: Behavioral: Cognitive tasks

INTERVENTIONS:
Behavioral: Cognitive tasks — MagnetoEncephaloGraphy (MEG) records

SUMMARY:
Depending on the point of view, different definitions of aging have been proposed. Thus, at the biological level, aging corresponds to a natural physiological process that leads to the progressive degeneration of cells and the slowing down of the vital functions of a living organism. More generally, aging is a multifactorial and multidimensional process that occurs at the cognitive, social, biological or psychological level.

The primary objective of this study is to evaluate the balance between activation (Task-Positive Network : TPN-Language, L, TPN-Verticality, V) and rest (Task-Negative Network : TNN) activity during normal aging, in two domains (language and posturo-spatial perception of verticality).

DETAILED DESCRIPTION:
From a cognitive point of view, although healthy older people become slower to analyze information, they remain just as accurate as young adults in performing different cognitive tasks. This necessarily implies compensation processes, with new cognitive strategies and a restructuring of the brain networks underlying these processes. These compensatory phenomena are known under the general name of neurocognitive reserve.

Specific functions such as language, visuospatial skills, motor control, posture, or memory, are affected in a very variable way among the elderly. This variability involves multiple cognitive profiles rather than just one form of aging. Indeed, healthy aging can be defined cognitively in two ways, as a homogeneous or rather heterogeneous process. According to the homogeneous hypothesis of aging, the behavioral, cognitive and brain-like manifestations are similar among the elderly, without differentiation between functions. In other words, according to this hypothesis, aging would affect all the elderly and cognitive processes in the same way. Conversely, according to the heterogeneous hypothesis, significant differences should be revealed between individuals and in the same individual according to different cognitive processes. This heterogeneity is explained by multiple factors (genetic, environmental, societal, educational, or lifestyle). If neuropsychological tests or behavioral experiments (and performance of the task) allow to identify rather easily the differences encountered among the elderly in terms of cognitive heterogeneity, this differential activity at the cerebral level is more difficult to highlight. Functional neuroimaging methods and techniques can provide a pathway for this purpose, to provide both spatial information (involved brain regions) and temporal information (dynamics of brain activation) when performing cognitive tasks or when the rest period.

In this context, the magnetoencephalography (MEG) method is a preferred technique that can provide all these types of information on brain activity. Two types of networks can therefore be recorded : task-positive network (TPN) activated when the participant is involved in a task (in this project, language and posture / verticality), and task-negative network (TNN) specific to the state of rest , represented by regions that are called "deactivated". These two networks will therefore be characterized in the study by the following parameters: (a) network: set of regions involved; (b) temporal dynamics of their activity, and (c) functional connectivity between the regions of TPN and TNN.

To answer the question of homogeneity vs. heterogeneity of cognitive cerebral aging, TPNs vs. TNN will be compared in a group of healthy young adults compared to a group of healthy elderly subjects. The comparison will be made for the three categories of parameters mentioned above (a-c).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers from 25 to 85 years old : young group (25-49 years) / aged group (50 to 85 years)
* Right-handed
* Signed informed consent
* French mother tongue
* Speaking fluent French
* Normal or corrected view
* Medical examination conducted prior to participation in the trial
* Registered in the French social security scheme

Exclusion Criteria:

* Contraindication to Magnetoencephalography (MEG) and/or Magnetic resonance imaging (MRI) : implanted material, claustrophobia,…
* Generally severe condition: cardiac, respiratory, hematological, kidney, liver, cancer
* Regular use of anxiolytics, sedatives, antidepressants, neuroleptics
* Psychiatric pathology characterized
* Alcohol ingestion before the exam
* All categories of protected persons (Pregnant or lactating women, persons subject to a legal protection measure, persons deprived of their liberty by judicial or administrative decision)
* Alcohol ingestion before the exam
* Participation in other ongoing clinical trial with exclusion period or in the previous week
* Score MINI MENTAL STATE EXAMINATION (MMSE) < 24

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Balance between activation (TPN-Language, L, TPN-Verticality, V) and rest (TNN) activity during normal aging, in two domains (language and posturo-spatial perception of verticality) recorded by magnetoencephalography (MEG) | 2 hours
  Evoked and continuous magnetic fields recorded during both cognitive tasks and during the rest period

SECONDARY OUTCOMES:
Correlation between neuropsychological scores and brain activation or functional connectivity parameters recorded by magnetoencephalography (MEG) depending on both domains studied | 1 hour
  Neuropsychological scores on tests for all participants :
  * frontal cognitive functioning
  * anxiety and/or depressive symptoms
  * executive functions
  * verbal intelligence
  * language
  Advanced analyses of cerebral activity as measured by MEG
  * frequency time analyses via spectral decomposition (induced brain rhythms)
  * functional and effective connectivity analysis through coherence, phase locking value, and Dynamic Causal Modelling measures

CONTACTS AND LOCATIONS:
Overall Officials: Monica BACIU, MD, PhD, Principal Investigator — CHUGA
Locations (1):
- CHUGA, Grenoble, France

REFERENCES:
- [Background] Hoyau E, Roux-Sibilon A, Boudiaf N, Pichat C, Cousin E, Krainik A, Jaillard A, Peyrin C, Baciu M. Aging modulates fronto-temporal cortical interactions during lexical production. A dynamic causal modeling study. Brain Lang. 2018 Sep;184:11-19. doi: 10.1016/j.bandl.2018.06.003. Epub 2018 Jun 15. PMID 29913316
- [Background] Baciu M, Boudiaf N, Cousin E, Perrone-Bertolotti M, Pichat C, Fournet N, Chainay H, Lamalle L, Krainik A. Functional MRI evidence for the decline of word retrieval and generation during normal aging. Age (Dordr). 2016 Feb;38(1):3. doi: 10.1007/s11357-015-9857-y. Epub 2015 Dec 28. PMID 26711670
- [Background] Boudiaf N, Laboissiere R, Cousin E, Fournet N, Krainik A, Baciu M. Behavioral evidence for a differential modulation of semantic processing and lexical production by aging: a full linear mixed-effects modeling approach. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2018 Jan;25(1):1-22. doi: 10.1080/13825585.2016.1257100. Epub 2016 Nov 24. PMID 27883290